CLINICAL TRIAL: NCT01156766
Title: Locking Plate Versus Pins for Surgical Treatment of Posteriorly Tilted Distal Radius Fracture
Brief Title: Metaphyseal Distal Radius Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Stryker SA (Industry); Polyclinique du Parc Rambot (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0077
Record Dates: First submitted 2010-07-02; First posted 2010-07-05 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Metaphyseal Radius Fractures (AO Type A2, A3, C1 et C2)
Keywords: Fracture; Radius; Osteosynthesis; Metaphyseal; Pinning; Locking anterior plate
MeSH Terms: conditions — Fractures, Bone

INTERVENTIONS:
Device: - locking anterior plate — The number of osteoporotic fractures, among which the fractures of the lower extremity of the radius (16 % of fractures seen in emergencies) is going to increase. Several surgical techniques are described in particular locking plates and intrafocal pinning techniques.
  The aim of the study is to compare (X-ray assessments and functional outcome) these two types of treatment by using a prospective, randomised multicentric analysis.

SUMMARY:
The number of osteoporotic fractures, among which the fractures of the lower extremity of the radius (16 % of fractures seen in emergencies) is going to increase. Several surgical techniques are described in particular locking plates and intrafocal pinning techniques.

The aim of the study is to compare (X-ray assessments and functional outcome) these two types of treatment by using a prospective, randomised multicentric analysis.

DETAILED DESCRIPTION:
Because an increasing number of elderly patient, the number of osteoporotic fractures, among which the fractures of the lower extremity of the radius (16 % of fractures seen in emergencies) is going to increase. Several surgical techniques exist of which in particular locking plates and intrafocal pinning.

The availability of new materials (locking plates with angular stability) seems to reduce the risks of osteosynthesis failure and seems to give more constant results: hawever, the price to pay is a more invasive technique and a superior cost. The rehabilitation seems also faster, allowing the possibility to get back the maximum of autonomy.

These clinical facts need of course to be validated.

ELIGIBILITY:
Inclusion Criteria:

* - metaphyseal inferior radius fractures (AO classification 23A2, 23A3, 23C1, 23C2)
* age 60 years or older

Exclusion Criteria:

* open fracture
* fractures AO classification: 23A1, 23C3, 23B1, 23B2, 23B3
* polytraumatized patient
* fractures older than 15 days
* infection of the operating site
* previous osseous disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
- X-ray assessments (preoperative, postoperative; 2 weeks, 5 weeks, 3, 6 and 12 mouths) | preoperative, postoperative; 2 weeks, 5 weeks, 3, 6 and 12 mouths

SECONDARY OUTCOMES:
PAIN score (2 weeks, 5 weeks, 3, 6 and 12 months) | 2 weeks, 5 weeks, 3, 6 and 12 months
Gartland, O'Brien, DASH and Euroquol EQ-5D scores (5 weeks, 3, 6 and 12 months) | 5 weeks, 3, 6 and 12 months
Grip and pinch strength (5 weeks, 3, 6 and 12 months) | 5 weeks, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane DESCAMPS, MD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France